CLINICAL TRIAL: NCT06322108
Title: Assessment of the Safety and Efficacy of Balstilimab in Combination With Botensilimab for the Treatment of Non-Small Cell Lung Cancer (IMMONC0008)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immune Oncology Research Institute (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMONC0008
Record Dates: First submitted 2024-02-28; First posted 2024-03-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Immunotherapy; Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Botensilimab + Balstilimab (Experimental): botensilimab 75 mg IV every 6 weeks (up to 4 doses) + balstilimab 240 mg IV every 2 weeks
  Interventions: Drug: Botensilimab + Balstilimab

INTERVENTIONS:
Drug: Botensilimab + Balstilimab — Botensilimab is a fragment crystallizable (Fc)-engineered human immunoglobulin G1 (IgG1) monoclonal antibody that targets cytotoxic T lymphocyte-associated protein 4 (CTLA-4). Balstilimab is a human monoclonal antibody that targets programmed cell death protein 1 (PD-1).
  Other Names: AGEN1181 + AGEN2034

SUMMARY:
The goal of this study is to see if the combination of immunotherapy agents botensilimab and balstilimab is safe and effective in participants with metastatic non-small cell lung cancer (NSCLC) as a first-line treatment.

DETAILED DESCRIPTION:
This is a single-arm, open-label phase II study to evaluate the safety and efficacy of the combination of botensilimab and balstilimab in participants with metastatic non-small cell lung cancer (NSCLC). The study will enroll participants with a histologically confirmed diagnosis of metastatic NSCLC and without targetable EGFR mutation or ALK rearrangement, while excluding those with untreated brain metastases or oligometastatic disease lacking targetable lesions.

The total estimated maximum time of study participation for each patient is approximately 49 months across 3 periods:

* Screening Period: approximately 28 days
* Treatment Period: up to 24 months, or until any criterion for stopping the study drug or withdrawal from the study occurs
* Follow-up Period: up to 24 months from last dose of study treatment for every patient who is alive

Study Duration

* Recruitment: 2 years
* Treatment: 2 years
* Follow-up: 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and IHC confirmed diagnosis of metastatic NSCLC which has not received any prior anticancer medicinal therapy for metastatic disease.
2. Negative for actionable EGFR mutations and ALK rearrangements.
3. Patients with recurrence after prior neoadjuvant or adjuvant chemotherapy or radiation therapy or immune checkpoint inhibitors for non-metastatic disease are eligible if recurrence occurred >6 months after the end of neoadjuvant or adjuvant treatment.
4. Documented informed consent of the participant and/or legally authorized representative
5. ≥ 18 years of age.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy ≥ 3 months.
8. Patients should have measurable metastatic disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and iRECIST guidelines.
9. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (within 7 days prior to day 1 of protocol therapy) (except subjects with Gilbert syndrome who must have a total bilirubin level of ≤3.0 × ULN).
10. Aspartate aminotransferase (AST) ≤ 2.5 x ULN, unless presence of liver metastases for which ≤ 5 x ULN is allowed (within 7 days prior to day 1 of protocol therapy).
11. Alanine aminotransferase (ALT) ≤ 2.5 x ULN, unless presence of liver metastases for which ≤ 5 x ULN is allowed (within 7 days prior to day 1 of protocol therapy).
12. Creatinine clearance ≥ 45 ml/min (within 7 days prior to day 1 of protocol therapy).
13. Alkaline phosphatase ≤ 3 x ULN (within 7 days prior to day 1 of protocol therapy).
14. Hemoglobin ≥ 9 g/dl (within 7 days prior to day 1 of protocol therapy).
15. Absolute neutrophil count (ANC) ≥ 1500/ul (within 7 days prior to day 1 of protocol therapy).
16. Platelets ≥ 100,000/mm^3 (within 7 days prior to day 1 of protocol therapy).
17. Albumin ≥ 3.0 g/dl (within 7 days prior to day 1 of protocol therapy).
18. Women of childbearing potential (WOCBP): negative serum pregnancy test (within 7 days prior to day 1 of protocol therapy)

    a) Females of non-childbearing potential are defined as: i. ≥ 50 years of age and has not had menses for greater than 1 year ii. Amenorrheic for ≥ 2 years without a hysterectomy and bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation iii. Status is post-hysterectomy, bilateral oophorectomy, or tubal ligation.
19. Male and female patients of reproductive potential must use effective methods of contraception (defined in Appendix A) or abstain from sexual activity for the course of the study through at least 90 days after the last dose of balstilimab and/or botensilimab
20. Is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Prior treatment with anti-CTLA-4 and anti-PD-(L)1 therapy. Note: Prior treatment with anti-PD-(L)1 therapy in the adjuvant setting is permitted if recurrence occurred >6 months after the end of adjuvant treatment.
2. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid dose ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
3. Prior allogeneic organ transplantation.
4. Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement.
5. Prior allergic reaction or hypersensitivity to any of the study drug components.
6. Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs.
7. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), serious uncontrolled cardiac arrhythmia requiring medication.

   a. QTcF (QTc interval corrected using Fridericia's formula) of > 480 ms.
8. Any persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] grade ≥ 2) from prior cancer therapy, excluding endocrinopathies stable on medication, stable neuropathy that is grade 2 or less, and alopecia.
9. Active brain metastases or leptomeningeal metastases with the following exceptions:

   a. Treated brain metastases require a) surgical resection, or b) stereotactic radiosurgery. Whole-brain radiation is not allowed. Subjects must have also discontinued steroid treatment 28 days prior to enrollment for the purpose of managing their brain metastases and they must be asymptomatic and radiologically stable ≥28 days before enrollment.
10. Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 730 days (or 2 years) prior to enrollment, i.e., subjects with a history of prior malignancy are eligible if treatment was completed at least 730 days (or 2 years) before enrollment and the subject has no evidence of disease. Subjects with history of prior early-stage basal/squamous cell skin cancer, low-risk prostate cancer eligible for active surveillance or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible.
11. Any evidence of current interstitial lung disease (ILD) or pneumonitis, or prior history of ILD or non-infectious pneumonitis requiring glucocorticoids.
12. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
13. History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
14. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine or booster < 7 days before C1D1. For vaccines requiring more than 1 dose, the full series should be completed prior to C1D1, when feasible. Booster shot not required but also must be administered > 7 days from C1D1 or > 7 days from future cycle on study.
15. Uncontrolled infection with human Immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required.
16. Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Subjects who are receiving or who have received anti-HBV therapy and have undetectable HBV DNA for at least 180 days prior to enrollment are eligible. Serological testing for HBV at screening is not required.
17. Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Subjects on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 180 days prior to enrollment. Serological testing for HCV at screening is not required.
18. Known active tuberculosis. Tuberculosis testing at screening is required.
19. Grade 3 or above neuropathy at the time of enrollment.
20. Dependence on total parenteral nutrition or intravenous hydration.
21. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
22. Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
12-Month Progression-Free Survival (PFS) | First dose to up to 12 months
  12-Month PFS is defined as the proportion of patients who remain alive and progression-free at 12 months from the first dose of investigational drug, where tumor progression is documented per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) and modified Response Evaluation Criteria in Solid Tumors version 1.1 for immune-based therapeutics (iRECIST) as assessed by investigator.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | First dose to up to 6 months
  ORR is defined as the proportion of subjects with a complete response (CR) or partial response (PR) per RECIST v1.1 and iRECIST, as assessed by investigator.
Disease Control Rate (DCR) | First dose to up to 6 months
  DCR is defined as the percentage of patients who have achieved complete response, partial response or stable disease per the RECIST v1.1 and iRECIST criteria.
Duration of Response (DOR) | First dose to up to 48 months
  DOR is defined as the time from initial objective radiographic response per RECIST v1.1 and iRECIST as assessed by investigator until the first documentation of progression or death, whichever occurs first.
Time to Next Treatment (TTNT) | First dose to up to 48 months
  TTNT is defined as the time from the first dose of investigational drug to the start date of a subsequent line of therapy.
Overall Survival (OS) Time | First dose to up to 48 months
  OS Time is defined as the time from the first dose of investigational drug until death to any cause.
Frequency, severity, and duration of treatment emergent adverse events (TEAEs) (Safety and tolerability) | First dose to up to 27 months
  Adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0), serious adverse events, AEs leading to treatment discontinuation or death.
Health-related quality of life (HRQoL) according to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | First dose to up to 25 months
  HRQoL is a patient-reported outcome (PRO) assessed using EORTC QLQ-C30.
Health-related quality of life according to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer (EORTC QLQ-LC29) | First dose to up to 25 months
  Patient-reported outcome assessed using EORTC QLQ-LC29
Health-related quality of life according to the 5 Level EuroQol 5 Dimension (EQ-5D-5L) questionnaire | First dose to up to 25 months
  Patient-reported outcome assessed using EQ-5D-5L
Correlation between baseline expression of PD-L1 by immunohistochemistry (IHC) and 12-month progression-free survival | First dose to up to 24 months
  PD-L1 expression at baseline will be assessed via immunohistochemistry and categorized into negative (<1%), low expression (1-49%), and high expression (>50%), and its correlation with 12-month progression-free survival will be investigated.
Correlation between baseline expression of PD-L1 by immunohistochemistry (IHC) and objective response rate | First dose to up to 24 months
  PD-L1 expression at baseline will be assessed via immunohistochemistry and categorized into negative (<1%), low expression (1-49%), and high expression (>50%), and its correlation with objective response rate will be investigated.
Correlation between existence of liver metastases on imaging at baseline and 12-month progression-free survival | First dose to up to 24 months
  Presence of liver metastases at baseline will be assessed via imaging and its correlation with 12-month progression-free survival will be investigated.
Correlation between existence of liver metastases on imaging at baseline and objective response rate | First dose to up to 24 months
  Presence of liver metastases at baseline will be assessed via imaging and its correlation with objective response rate will be investigated.
Level of circulating tumor DNA (ctDNA) at baseline and at different time points after start of treatment | First dose to up to 24 months
  Level of ctDNA will be measured at screening, after start of treatment at 2 weeks, 4 weeks, 8 weeks, and at treatment discontinuation/disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Gevorg Tamamyan, MD, PhD, DSc, Study Director — Immune Oncology Research Institute; Samvel Bardakhchyan, MD, PhD, Study Chair — Immune Oncology Research Institute; Samvel Bardakhchyan, MD, PhD, Principal Investigator — Immune Oncology Research Institute
Locations (1):
- Hematology Center named after prof. R. Yeolyan, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No